CLINICAL TRIAL: NCT01059643
Title: A Phase 2 Indication Identification Study of LY2523355 in Patients With Ovarian, Non-Small Cell Lung, Prostate, Colorectal, Gastroesophageal Cancers, and Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Study in Ovarian, Non-Small Cell Lung, Prostate, Colorectal, Gastroesophageal Cancers, and Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12848; I1Y-MC-JFBF (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-01-11; First posted 2010-02-01 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer; Non Small Cell Lung Cancer; Prostate Cancer; Colorectal Cancer; Gastric Cancer; Esophageal Cancer; Cancer of Head and Neck
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms | interventions — litronesib; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2523355 (Experimental)
  Interventions: Drug: LY2523355; Drug: pegfilgrastim

INTERVENTIONS:
Drug: LY2523355 — Dose determined by participant body surface area: 5 milligrams/square meter(mg/m²) or 6 mg/m², administered intravenously as a 1-hour infusion on Days 1, 2 and 3 of a 21 day cycle; for up to 2 cycles (4 cycles for prostate cancer patients). Additional cycles administered based on patient response assessment.
Drug: pegfilgrastim — 6 milligrams (mg), administered subcutaneously approximately 24 hours after third dose of LY2523355 on Day 4 of each 21-day cycle, for up to 2 cycles of LY2523355 administration (4 cycles for prostate cancer patients). Additional cycles of LY2523355 administered based on patient response assessment.

SUMMARY:
The purpose of the study is to estimate the rate of response for patients with ovarian, non-small cell lung, prostate, colorectal, gastroesophageal, and head and neck cancers who are administered LY2523355.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian, non-small cell lung, prostate, colorectal, gastroesophageal cancer (adenocarcinoma of the esophageal cancer, stomach, or gastroesophageal junction), or squamous cell cancer of the head and neck
* Have measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines (except prostate cancer participants)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Are willing to follow study procedures for the duration of the study
* Are willing to use an approved contraceptive method during treatment and for 3 months after discontinuation of study treatment

Exclusion Criteria:

* Have a serious preexisting medical condition that would preclude participation in the study
* Are pregnant or lactating
* Have received treatment within 28 days of first dose of LY2523355 with a drug that has not received regulatory approval for any indication
* Have symptomatic, untreated, or uncontrolled central nervous system (CNS) metastases
* Have a second active primary malignancy or a history of a second malignancy requiring cytotoxic therapy
* Have QTc interval greater than 470 millisecond (msec) or intraventricular conduction delay (IVCD) with QRS greater than 120 msec on screening electrocardiogram (ECG)
* Have active symptomatic fungal, bacterial, and/or known viral infection including active human immunodeficiency virus (HIV) or viral (A, B, C) hepatitis
* Participants with pneumonia, evidence of obstructive pneumonitis, other respiratory infections, or infection from other sources are to be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1- 317-615-4559 Mon - Fri 9 AM to 5 PM (Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jonesboro, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdosta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Post Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westwood, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wichita, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Germantown, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corpus Christi, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who received at least one dose of study drug in both Cycle 1 and Cycle 2 or to have progressed or died on or before study Day 42 were considered to be completed.
Groups:
- LY2523355: LY2523355: Dose determined by participant's body surface area: 5 milligrams/square meter(mg/m²) or 6 mg/m², administered intravenously as a 1-hour infusion on Days 1, 2 and 3 of a 21-day cycle for up to 2 cycles (4 cycles for prostate cancer participants). Additional cycles administered based on participant response assessment.
  Pegfilgrastim: 6 milligrams (mg), administered subcutaneously approximately 24 hours after third dose of LY2523355 on Day 4 of each 21-day cycle, for up to 2 cycles of LY2523355 administration (4 cycles for prostate cancer participants). Additional cycles of LY2523355 administered based on participant response assessment.
Period: Overall Study
Arm/Group | LY2523355
Started | 103
Received at Least 1 Dose of Study Drug | 103
Completed | 97
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY2523355: LY2523355: Dose determined by participant body surface area: 5 milligrams/square meter(mg/m²) or 6 mg/m², administered intravenously as a one hour infusion on Days 1, 2 and 3 of a 21 day cycle for up to 2 cycles (4 cycles for prostate cancer participants). Additional cycles administered based on participant response assessment.
  Pegfilgrastim: 6 milligrams (mg), administered subcutaneously approximately 24 hours after third dose of LY2523355 on Day 4 of each 21-day cycle, for up to 2 cycles of LY2523355 administration (4 cycles for prostate cancer participants). Additional cycles of LY2523355 administered based on participant response assessment.
Arm/Group | LY2523355
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 101
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 93
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 103
Tumor Type [Number; unit: participants]
  Colorectal Cancer | 17
  Gastroesophageal Cancer | 13
  Non-Small Cell Lung Cancer | 29
  Ovarian Cancer | 13
  Prostate Cancer | 18
  Squamous Cell Carcinoma of the Head and Neck | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response (CR) or Partial Response (PR)
Description: The percentage of participants who achieved a best response of either CR or PR, as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions. PR was defined as at least a 30% decrease in sum of longest diameter of target lesions and for prostate cancer PR was defined as a ≥50% decrease in baseline prostate-specific antigen (PSA) value that was confirmed with a second value ≥3 weeks later. Progressive Disease (PD) was defined as at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase over nadir. Percentage is calculated as a total number of participants with CR or PR divided by the total number of participants treated multiplied by 100.
Time Frame: Baseline until progressive disease up to 36 weeks post-baseline
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY2523355
Number analyzed (Participants) | 103
percentage of participants
  Colorectal Cancer: number analyzed (Participants) | 17
  Colorectal Cancer | 0 [0.0 to 17.1]
  Gastroesophageal Cancer: number analyzed (Participants) | 13
  Gastroesophageal Cancer | 0 [0.0 to 22.1]
  Non-Small Cell Lung Cancer: number analyzed (Participants) | 29
  Non-Small Cell Lung Cancer | 0 [0.0 to 10.9]
  Ovarian Cancer: number analyzed (Participants) | 13
  Ovarian Cancer | 0 [0.0 to 20.6]
  Prostate Cancer: number analyzed (Participants) | 18
  Prostate Cancer | 0 [0.0 to 16.2]
  Squamous Cell Carcinoma of Head and Neck: number analyzed (Participants) | 13
  Squamous Cell Carcinoma of Head and Neck | 0 [0.0 to 25.9]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from date of first dose to the first observation of disease progression or death due to any cause. Progressive Disease (PD) was defined as at least 20% increase in sum of longest diameter of target lesions and minimum 5 millimeter (mm) increase over nadir. For participants who were not known to have died or to have progressed as of the data inclusion cutoff date, PFS were censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systemic anticancer therapy.
Time Frame: Date of enrollment to progressive disease or death due to any cause up to 36 weeks post-enrollment
Population: All enrolled participants who received at least 1 dose of study drug. Percentage (%) of participants censored were colorectal cancer 5.9%; gastroesophageal cancer 0.0%, non-small cell lung cancer 3.4%, ovarian cancer 15.4%, prostate cancer 16.7%, and squamous cell carcinoma of the head and neck 15.4%.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | LY2523355
Number analyzed (Participants) | 103
months
  Colorectal Cancer: number analyzed (Participants) | 17
  Colorectal Cancer | 1.30 [1.28 to 2.69]
  Gastroesophageal Cancer: number analyzed (Participants) | 13
  Gastroesophageal Cancer | 1.25 [0.62 to 1.51]
  Non-Small Cell Lung Cancer: number analyzed (Participants) | 29
  Non-Small Cell Lung Cancer | 1.31 [1.28 to 1.91]
  Ovarian Cancer: number analyzed (Participants) | 13
  Ovarian Cancer | 1.31 [1.18 to 2.10]
  Prostate Cancer: number analyzed (Participants) | 18
  Prostate Cancer | 2.30 [1.45 to 2.66]
  Squamous Cell Carcinoma of Head and Neck: number analyzed (Participants) | 13
  Squamous Cell Carcinoma of Head and Neck | 1.51 [0.72 to 2.76]

3. Secondary Outcome: Percentage of Participants Who Achieved a Best Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD)
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions. PR was defined as at least a 30% decrease in sum of longest diameter of target lesions and for prostate cancer PR was defined as a ≥50% decrease in baseline prostate-specific antigen (PSA) value that was confirmed with a second value ≥3 weeks later. Progressive Disease (PD) was defined as at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase over nadir. SD was defined as small changes that did not meet above criteria.
Time Frame: Baseline until progressive disease up to 36 weeks post-baseline
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | LY2523355
Number analyzed (Participants) | 103
percentage of participants
  Colorectal Cancer: number analyzed (Participants) | 17
  Colorectal Cancer | 37.5 [17.8 to 60.9]
  Gastroesophageal Cancer: number analyzed (Participants) | 13
  Gastroesophageal Cancer | 16.7 [3.0 to 43.8]
  Non-Small Cell Lung Cancer: number analyzed (Participants) | 29
  Non-Small Cell Lung Cancer | 38.5 [22.6 to 56.4]
  Ovarian Cancer: number analyzed (Participants) | 13
  Ovarian Cancer | 30.8 [11.3 to 57.3]
  Prostate Cancer: number analyzed (Participants) | 18
  Prostate Cancer | 47.1 [26.0 to 68.9]
  Squamous Cell Carcinoma of Head and Neck: number analyzed (Participants) | 13
  Squamous Cell Carcinoma of Head and Neck | 50.0 [22.2 to 77.8]

4. Secondary Outcome: Tumor Marker Values as Relevant to Specific Tumor Types at Baseline
Description: The number of participants with colorectal cancer (CRC), gastroesophageal cancer (GE), non-small cell lung cancer (NSCLC), ovarian cancer, prostate cancer or squamous cell carcinoma of head and neck (SCCHN) who had marker/molecular diagnostics performed prior to study entry to determine the mutation status of cancer genes: APC, BRAF, BRCA1, BRCA2, HRAS and KRAS and the presence of Human Papillovirus (HPV) and Epstein Barr viruses (EBV). Mutation/virus status was defined as: positive (mutation/virus present), negative (mutation/virus not present), unknown (mutation/virus status unknown), or not done (mutation/virus status was not done).
Time Frame: Baseline
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2523355
Number analyzed (Participants) | 103
Participants
  CRC-BRAF Mutation, Negative: number analyzed (Participants) | 17
  CRC-BRAF Mutation, Negative | 2
  CRC-BRAF Mutation, Not Done/Unknown: number analyzed (Participants) | 17
  CRC-BRAF Mutation, Not Done/Unknown | 15
  CRC-KRAS Mutation, Positive: number analyzed (Participants) | 17
  CRC-KRAS Mutation, Positive | 9
  CRC-KRAS Mutation, Negative: number analyzed (Participants) | 17
  CRC-KRAS Mutation, Negative | 7
  CRC-KRAS Mutation, Not Done: number analyzed (Participants) | 17
  CRC-KRAS Mutation, Not Done | 1
  GE-KRAS Mutation, Negative: number analyzed (Participants) | 13
  GE-KRAS Mutation, Negative | 1
  GE-KRAS Mutation, Not Done/Unknown: number analyzed (Participants) | 13
  GE-KRAS Mutation, Not Done/Unknown | 12
  NSCLC-KRAS Mutation, Positive: number analyzed (Participants) | 29
  NSCLC-KRAS Mutation, Positive | 3
  NSCLC-KRAS Mutation, Negative: number analyzed (Participants) | 29
  NSCLC-KRAS Mutation, Negative | 5
  NSCLC-KRAS Mutation, Not Done/Unknown: number analyzed (Participants) | 29
  NSCLC-KRAS Mutation, Not Done/Unknown | 21
  Ovarian-BRCA1 Mutation, Negative: number analyzed (Participants) | 13
  Ovarian-BRCA1 Mutation, Negative | 3
  Ovarian-BRCA1 Mutation, Not Done/Unknown: number analyzed (Participants) | 13
  Ovarian-BRCA1 Mutation, Not Done/Unknown | 10
  Ovarian-BRCA2 Mutation, Negative: number analyzed (Participants) | 13
  Ovarian-BRCA2 Mutation, Negative | 3
  Ovarian-BRCA2 Mutation, Not Done/Unknown: number analyzed (Participants) | 13
  Ovarian-BRCA2 Mutation, Not Done/Unknown | 10
  SCCHN-APC Mutation, Negative: number analyzed (Participants) | 13
  SCCHN-APC Mutation, Negative | 1
  SCCHN-APC Mutation, Not Done/Unknown: number analyzed (Participants) | 13
  SCCHN-APC Mutation, Not Done/Unknown | 12
  SCCHN-HPV (HPV-31 Positive) Mutation: number analyzed (Participants) | 13
  SCCHN-HPV (HPV-31 Positive) Mutation | 1
  SCCHN-HPV Mutation, Not Done/Unknown: number analyzed (Participants) | 13
  SCCHN-HPV Mutation, Not Done/Unknown | 12

5. Secondary Outcome: Change in Tumor Size at Smallest Size (Best Response)
Description: The percent change in tumor size at its smallest size. The sum of diameters of target lesions was determined at each tumor assessment. The percent change is the smallest post-baseline sum divided by the baseline (pre-treatment) sum, multiplied by 100.
Time Frame: Baseline until cycle with maximum change from baseline up to 36 weeks
Population: All enrolled participants who received at least 1 dose of study drug with results at baseline and at time of best response.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | LY2523355
Number analyzed (Participants) | 73
percentage of change
  Colorectal Cancer: number analyzed (Participants) | 16
  Colorectal Cancer | 15.4 (17.12)
  Gastroesophageal Cancer: number analyzed (Participants) | 10
  Gastroesophageal Cancer | 29.0 (70.00)
  Non-Small Cell Lung Cancer: number analyzed (Participants) | 23
  Non-Small Cell Lung Cancer | 21.9 (48.69)
  Ovarian Cancer: number analyzed (Participants) | 11
  Ovarian Cancer | 22.1 (31.40)
  Prostate Cancer: number analyzed (Participants) | 5
  Prostate Cancer | 12.2 (15.91)
  Squamous Cell Carcinoma of Head and Neck: number analyzed (Participants) | 8
  Squamous Cell Carcinoma of Head and Neck | 3.9 (30.67)

6. Secondary Outcome: Pharmacokinetics, Maximum Plasma Concentration (Cmax) of LY2523355 and Metabolite LSN2546307
Description: Plasma Cmax following daily doses of LY2523355 on Days 1, 2, and 3 of Cycle 1 (21-day cycle).
Time Frame: Day 3 of Cycle 1 (21-day cycle)
Population: All enrolled participants who received at least 1 dose of study drug with Cmax measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 5 mg/m² LY2523355: LY2523355: 5 milligrams/square meter/day (mg/m²/day) administered intravenously as a 1-hour infusion on Days 1, 2, and 3 + pegfilgrastim on Day 4 of each 21-day cycle.
- 6 mg/m² LY253355: LY2523355: 6 mg/m²/day administered intravenously as a one hour infusion on Days 1, 2, and 3 + pegfilgrastim on Day 4 of each 21-day cycle.
Arm/Group | 5 mg/m² LY2523355 | 6 mg/m² LY253355
Number analyzed (Participants) | 65 | 31
nanograms per milliliter (ng/mL)
  LY2523355 | 125 (79) | 124 (67)
  LSN2546307 | 5.0 (51) | 5.3 (52)

7. Secondary Outcome: Pharmacokinetics, Intracycle Accumulation Ratio (Ra) of LY2523355
Description: Intracycle Ra of LY2523355 is the ratio of LY2523355 maximum plasma concentration (Cmax) on Day 3 of Cycle 1 to the Cmax of LY2523355 on Day 1 of Cycle 1 following daily doses of LY2523355 on Days 1, 2 and 3 of Cycle 1 (21-day cycle) at each dose level.
Time Frame: Day 1 and Day 3 of Cycle 1 (21-day cycle)
Population: All enrolled participants who received at least 1 dose of study drug with Ra measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Groups:
- 5 mg/m²LY2523355: LY2523355: 5 milligrams/square meter/day (mg/m²/day) administered intravenously as a 1-hour infusion on Days 1, 2, and 3 + pegfilgrastim on Day 4 of each 21-day cycle.
Arm/Group | 5 mg/m²LY2523355 | 6 mg/m² LY253355
Number analyzed (Participants) | 65 | 28
ratio | 1.02 (87) | 1.08 (61)

8. Other Pre Specified Outcome: Number of Participants Who Died Due to Unknown Causes During the 30-Day Post-Study Treatment Follow-Up
Time Frame: End of study treatment up to 30-days post-study treatment discontinuation
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2523355
Number analyzed (Participants) | 103
Participants | 5

ADVERSE EVENTS:
Description: Deaths due to (d/t) PD not considered AEs and reported in Participant Flow for those who died during study treatment. Deaths d/t unknown cause in the 30-day post-study treatment follow-up (PSTF) reported in Other Pre-Specified Outcome Measure. One death (unknown cause) in PSTF recorded by investigator as an SAE included in SAE summary as "Death".
Groups:
- LY2523355: LY2523355: Dose determined by participant's body surface area: 5 milligrams/meter squared (mg/m²) or 6 mg/m², administered intravenously on days 1, 2, 3 of a 21 day cycle; for up to 2 cycles (4 cycles for prostate cancer participants). Additional cycles administered based on participant response assessment.
  Pegfilgrastim: 6 milligrams (mg), administered subcutaneously 24 hours after third dose of LY2523355 on day 4 of each 21-day cycle, for up to 2 cycles of LY2523355 administration (4 cycles for prostate cancer participants). Additional cycles of LY2523355 administered based on participant response assessment.
Arm/Group | LY2523355
Serious Adverse Events (participants affected / at risk) | 39/103
Other Adverse Events (participants affected / at risk) | 102/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2523355 (N=103)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (6)
Pericardial effusion (Cardiac disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 5 (6)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Rectal abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4) — 1 event resulted in death
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) — Event resulted in death
Mental status changes (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) — 1 event resulted in death
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2523355 (N=103)
Anaemia (Blood and lymphatic system disorders) | 33 (52)
Neutropenia (Blood and lymphatic system disorders) | 21 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (18)
Abdominal pain (Gastrointestinal disorders) | 11 (12)
Constipation (Gastrointestinal disorders) | 24 (25)
Diarrhoea (Gastrointestinal disorders) | 18 (22)
Dysphagia (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 35 (38)
Oral pain (Gastrointestinal disorders) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 14 (15)
Vomiting (Gastrointestinal disorders) | 18 (19)
Asthenia (General disorders) | 6 (7)
Fatigue (General disorders) | 45 (54)
Mucosal inflammation (General disorders) | 19 (22)
Oedema peripheral (General disorders) | 10 (13)
Pyrexia (General disorders) | 9 (11)
Urinary tract infection (Infections and infestations) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 8 (8)
Blood creatinine increased (Investigations) | 7 (7)
Weight decreased (Investigations) | 10 (10)
White blood cell count decreased (Investigations) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 26 (29)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Dizziness (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 10 (10)
Anxiety (Psychiatric disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12)
Hypotension (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days